CLINICAL TRIAL: NCT06514768
Title: Early Exploratory Clinical Study on the Safety, Tolerability and Preliminary Efficacy of JY231 Injection in the Treatment of Acute B Lymphoblastic Leukemia
Brief Title: JY231 (JY231) Injection for the Treatment of B-cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-23-006
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia (B-ALL)
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY231 injection for the treatment of B-cell acute lymphoblastic leukemia (B-ALL) (Experimental)
  Interventions: Biological: JY231

INTERVENTIONS:
Biological: JY231 — Infusion of JY231 Injection by dose of 1-10×10^6 Transduction Units (TU)/kg、1-5×10^7 TU/kg、5-10 ×10^7 TU/kg. Administration method: intravenous infusion、Splenic artery infusion、Lymph node infusion; Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion (PI evaluation is required)

SUMMARY:
Early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of B-cell acute lymphoblastic leukemia (B-ALL)

ELIGIBILITY:
Inclusion Criteria:

1. up to 75 years (Child, Adult) , either sex；
2. Bone marrow cell morphology examination showed the proportion of primitive and immature lymphocytes in the bone marrow is >5%, or the bone marrow MRD analysis comfirmed as B-ALL.
3. Flow cytometry or histology confirmed positive expression of cluster of differentiation 19 (CD19);
4. According to the researcher's assessment, the expected survival period is greater than 3 months;
5. Eastern Cooperative Oncology Group (ECOG) physical condition score ≤ 3;
6. The patient has good liver, kidney, heart, and lung functions: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal(ULN), which can be relaxed to ≤ 5 × ULN for patients with liver invasion; Total serum bilirubin < 34 μ Mol/L; Creatinine clearance rate>30 mL/min; Cardiac ejection fraction (EF) ≥ 40%, without pericardial effusion and significant arrhythmia; Indoor oxygen saturation (SpO2) ≥ 92%;
7. Peripheral blood lymphocyte absolute count: absolute lymphocyte count (ALC) ≥ 0.5E9/L, blood platelet (PLT) > 30E9/L, Hb > 80g/L, with a single venous access and no other contraindications for blood cell separation;
8. MRI examination showed no active malignant cells in the cerebrospinal fluid, no brain metastases, or no central nervous system leukemia;
9. Individuals with fertility must agree to the use of efficient contraceptive methods;
10. The subject or their legal guardian can understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women, as well as women with pregnancy plans within six months;
2. Virological tests of hepatitis B, hepatitis C, AIDS, syphilis and cytomegalovirus were positive;
3. Having a history of other tumors (excluding skin or cervical carcinoma in situ cured by root therapy and without evidence of disease activity);
4. Previously received treatment targeting CD19;
5. Received autologous hematopoietic stem cell transplantation within 6 weeks;
6. The presence of uncontrollable active bacterial or fungal infections;
7. Allergies to research related drugs or cellular components;
8. Active autoimmune diseases exist;
9. Patients with unstable or active ulcers or gastrointestinal bleeding currently present;
10. Individuals with mental or psychological disorders who cannot cooperate with treatment and efficacy evaluation;
11. Received other experimental drug treatments within the past 3 months;
12. Existence of grade II-IV acute graft versus-host disease (GVHD) or widespread chronic GVHD;
13. Researchers believe that other reasons are not suitable for clinical trial participants.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
MTD | Up to 28 days after infusion
  MTD will be determined based on DLTs observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | At 2,4,8 and 12 weeks after infusion
  Overall Response Rate (ORR) is defined as the proportion of subjects achieving complete remission (CR) and complete remission with incomplete hematological recovery (CRi).
Best Overall Response | Up to 24 weeks after infusion
  The optimal degree of disease status improvement achieved by the patient over the course of the entire clinical trial or treatment period.
Duration of remission (DOR) | Up to 2 years after infusion
  Duration of remission (DOR) is the time from the first detection of CR or PR to the discovery of PD.
Time To Progression (TTP) | Up to 2 years after infusion
  The duration from the initiation of treatment until the first occurrence of objective disease progression.
Progression-free survival (PFS) | Up to 2 years after infusion
  Progression-free survival (PFS) is the time between the time a patient with tumor disease receives treatment and the time between the observation of disease progression or death from any cause.
Overall survival (OS) | Up to 2 years after infusion
  Overall survival (OS) is the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th HJointLogistics, Kunming, Yunnan, China